CLINICAL TRIAL: NCT05728346
Title: A Single-arm Clinical Trial Evaluating the Efficacy and Safety of Pulp Regeneration Induced by SHED Polymerization in Patients With Pulp Necrosis of Permanent Teeth
Brief Title: The Efficacy and Safety of Pulp Regeneration Induced by SHED Polymerization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Xueli Mao, Chief physician, Fifth Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xueli Mao
Record Dates: First submitted 2023-01-30; First posted 2023-02-15 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Pulp Necroses
Keywords: pulp necrosis; pulp regeneration
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm (Experimental)
  Interventions: Drug: Allogeneic human pulp mesenchymal stem cells mixed with hyaluronic acid polymers

INTERVENTIONS:
Drug: Allogeneic human pulp mesenchymal stem cells mixed with hyaluronic acid polymers — stem cells from human exfoliated deciduous teeth (SHED) mixed with hyaluronic acid polymers

SUMMARY:
Dental pulp necrosis is one of the most common pathological conditions that results in tooth loss. However, regeneration of functional dental pulp has proved difficult. Therefore, the investigators conduct a single-arm study to evaluate the efficacy and safety of pulp regeneration induced by SHED mixed with hyaluronic acid polymerization in patients with pulp necrosis of permanent teeth.

DETAILED DESCRIPTION:
This study is a single-center, prospective, single-arm study to evaluate the efficacy and safety of pulp regeneration induced by SHED mixed with hyaluronic acid polymerization in patients with pulp necrosis of permanent teeth. This study plans to include 30 subjects from the Department of Stomatology of the Fifth Affiliated Hospital of Guangzhou Medical University. All participants in this study will receive stem cells from human exfoliated deciduous teeth (SHED) mixed with hyaluronic acid polymers after the preparation and disinfection of the root canal of the affected teeth. All participants will undergo screening and baseline visits. After surgery, the participants will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 45 years
* Patients with pulp necrosis of a single canal permanent tooth due to trauma or caries
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with pulp necrosis caused by severe trauma to the tooth, such as crown root fracture, tooth root fracture, tooth displacement, etc
* Patients with calcification of the apical foramen at the root of the tooth
* History of hereditary disorders of abnormal tooth development
* Dental occlusal trauma, bruxism, malocclusion
* Bad oral habits (sticking out the tongue, biting lips, biting nails, sucking fingers, etc.)
* Presence of uncontrollable pathological processes in the oral cavity (presence of acute advanced diseases in the oral cavity)
* Malnutrition (serum albumin concentration<2 g/dl)
* Patients with history of other systemic, communicable or hereditary diseases have been diagnosed
* Pregnant, nursing, planning to become pregnant
* The investigators determined that the patient was not suitable for the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of pulp vitality | 1、3、6、12、18、24 months
  Change in pulpal vitality will be assessed through pulpal response to sensitivity tests (cold, hot and electrical test) in affected tooth.

SECONDARY OUTCOMES:
Blood flow in the root of tooth | 1、3、6、12、18、24 months
  Detection rate of blood flow in the root canal of the affected tooth by laser doppler flowmetry.